CLINICAL TRIAL: NCT00291811
Title: Compassionate Use Protocol for the Use of AMD3100 to Mobilize Peripheral Blood Stem Cells for Collection and Transplantation
Brief Title: Access Program for Use of AMD3100 to Increase Peripheral Blood Stem Cells for Transplantation in Patients Who Have Failed Standard Therapy Stem Cell Mobilization
Acronym: CUP
Status: Approved for marketing | Type: Expanded Access
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: AMD3100-CUP001
Record Dates: First submitted 2006-02-13; First posted 2006-02-15 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Autologous Stem Cell Transplant
Keywords: AMD3100; G-CSF
MeSH Terms: interventions — plerixafor; Granulocyte Colony-Stimulating Factor

INTERVENTIONS:
Drug: AMD3100 + G-CSF — Subcutaneous injection of 240 mcg/kg on the evening prior to each apheresis session
  Other Names: Plerixafor(injection)

SUMMARY:
The purpose of this program is to provide access to AMD3100 for patients who would benefit from an autologous stem cell transplant but who have either previously failed to collect enough cells for transplant following standard therapy or are not considered by their physician to have a reasonable chance of collecting enough cells for transplant.

DETAILED DESCRIPTION:
The purpose of this program is to provide access to AMD3100 for patients who would benefit from an autologous stem cell transplant but who have either previously failed to collect enough cells for transplant following standard therapy or are not considered by their physician to have a reasonable chance of collecting enough cells for transplant.

Compassionate use is a way to provide experimental treatment to a patient who is not eligible to receive that therapy in a clinical trial, but who has a serious or life-threatening illness for which other treatments are not available.

Peripheral blood stem cells are obtained by apheresis following a stem cell mobilization regimen. The standard of care regimen for stem cell mobilization includes a growth factor, G-CSF. AMD3100 is given in addition to G-CSF prior to each apheresis session. If enough peripheral blood stem cells for transplant are collected, the patient is treated with high dose chemotherapy in preparation for transplant and is transplanted with cells obtained from the AMD3100 and G-CSF regimen. Patients are followed for safety and transplant outcomes for up to 12 months after transplant.

ELIGIBILITY:
Inclusion Criteria:

* Patient is eligible for autologous transplant
* Patient has failed previous conventional therapies for stem cell collection, or is not considered by the physician to have a reasonable chance of collecting enough cells for transplant
* Patient has Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Patient has recovered from all acute toxic effects of prior chemotherapy
* Patient has white blood cell count greater than 2.5 x 10^9 cells/L
* Patient has absolute neutrophil count (ANC) greater than 1.5 x 10^9 cells/L
* Patient has platelet count greater than 85 x 10^9 cells/L
* Patient has serum creatinine less than or equal to 1.5 mg/dL
* Patient has creatinine clearance greater than 60 mL/min
* Patient has liver function tests less than 2x upper limit of normal
* Patient has left ventricle ejection fraction greater than 45%
* Patient has forced expiratory volume in 1 second (FEV1) greater than 60% of predicted or diffusing capacity of lung carbon monoxide (DLCO) and greater than or equal to 45% of predicted
* Patient has no active infection of hepatitis B or C
* Patient is negative for HIV
* Patient has signed informed consent
* Women of child bearing potential agree to use an approved form of contraception

Exclusion Criteria:

* Patients with leukemia (Note: Patients with multiple myeloma must be evaluated for plasma cells or blasts within 24 hours prior to the first dose of AMD3100)
* Patient has an existing condition which, in the view of the Investigator, renders the patient at high risk from treatment complications
* Patient has a residual acute medical condition resulting from prior chemotherapy
* Patient has brain metastases or carcinomatous meningitis
* Patient has an acute infection
* Patient has a fever (temperature greater than 38 degrees C/100.4 degrees F)
* Patient has hypercalcaemia greater than 1 mg/dL above the upper limit of normal
* Female patient has positive pregnancy test
* Female patient is lactating
* Patient is of child-bearing potential and is unwilling to use adequate birth control
* Patients with actual body weight exceeding 175% of their ideal body weight
* Patients who previously received experimental therapy within 4 weeks of enrolling in this protocol or who are currently enrolled in another experimental protocol
* Patients who experience a deterioration in health between the time of enrollment and transplant (such that they no longer meet entry criteria) may be removed from study at the discretion of the treating physician, principal Investigator, or Sponsor

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-10

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company

REFERENCES:
- [Derived] Deol A, Abrams J, Masood A, Al-Kadhimi Z, Abidi MH, Ayash L, Lum LG, Ratanatharathorn V, Uberti JP. Long-term follow up of patients proceeding to transplant using plerixafor mobilized stem cells and incidence of secondary myelodysplastic syndrome/AML. Bone Marrow Transplant. 2013 Aug;48(8):1112-6. doi: 10.1038/bmt.2013.10. Epub 2013 Mar 11. PMID 23474805